CLINICAL TRIAL: NCT07383545
Title: The Effect of Awareness Training on Peer Bullying Applied to Adolescents on Peer Bullying, Empathy, and Sympathy Levels
Brief Title: The Effect of Awareness Training on Peer Bullying
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Alime Selçuk Tosun, Associate Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023/82
Record Dates: First submitted 2026-01-25; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Bullying and Victimization
Keywords: Adolescent; Peer bullying; Victimization; Empathy; Sympathy
MeSH Terms: conditions — Bullying

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Awareness training on peer bullying (Experimental): Participants in the intervention group received a peer bullying awareness training program consisting of five sessions, delivered once per week. Each session lasted 40-45 minutes and was delivered in small groups. The program focused on increasing awareness of peer bullying, reducing bullying and victimization behaviors, and enhancing empathy and sympathy skills.
  Interventions: Behavioral: Awareness training on peer bullying
- Usual Care Control Group (No Intervention): Participants in the control group did not receive any intervention and continued with their usual school routine during the study period.

INTERVENTIONS:
Behavioral: Awareness training on peer bullying — Participants in the intervention group received a peer bullying awareness training program consisting of five sessions, delivered once per week. Each session lasted 40-45 minutes and was delivered in small groups. The program focused on increasing awareness of peer bullying, reducing bullying and victimization behaviors, and enhancing empathy and sympathy skills.
  Arms: Awareness training on peer bullying

SUMMARY:
This study examined the effect of awareness training on peer bullying, victimization, empathy, and sympathy levels in adolescents. A total of 64 students were randomly assigned to an intervention group or control group. The intervention group received five sessions of peer bullying awareness training, while the control group received no intervention. Data were collected using the Peer Bullying Identification Scale and the Empathy and Sympathy Scale.

ELIGIBILITY:
Inclusion Criteria:

* Being enrolled in the 9th grade
* Scoring 54 or higher on the Peer Bullying Identification Scale - Adolescent Form
* Willingness to participate and providing informed consent

Exclusion Criteria:

* Previous participation in a similar peer bullying or awareness training program
* Being a foreign national student due to insufficient proficiency in Turkish language comprehension and expression
* Missing two or more sessions of the peer bullying awareness training program

Ages: 14 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Peer Bullying Identification Scale - Adolescent Form | At baseline and one week after completion of the intervention
  Peer bullying and victimization levels will be assessed using the Peer Bullying Identification Scale - Adolescent Form. The minimum score that can be obtained from the bully and victim subscales of the scale is 53, and the maximum score is 265. As the score obtained from the scale increases, the level of being a bully and a victim also increases.

SECONDARY OUTCOMES:
Empathy and Sympathy Scale in Adolescents | At baseline and one week after completion of the intervention
  Empathy and sympathy levels will be measured using the Empathy and Sympathy Scale in Adolescents, which includes cognitive empathy, emotional empathy, and sympathy subscales. The minimum score that can be obtained from the scale is 12, and the maximum score is 60. The scale score is calculated by taking the mean of the item scores. A high score obtained from the scale indicates a high level of empathy or sympathy, whereas a low score indicates a low level of empathy or sympathy.

CONTACTS AND LOCATIONS:
Overall Officials: Alime Selçuk Tosun, Principal Investigator — Selcuk University, Faculty of Nursing
Locations (1):
- Karaman Bifa Anatolian High School, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to ethical restrictions and the need to protect participant confidentiality, as the study involves adolescent participants.

REFERENCES:
- [Background] Seyhan Sahin S, Ayaz-Alkaya S. The effect of motivational interviewing on peer bullying and cyberbullying in adolescents: A randomized controlled trial. J Nurs Scholarsh. 2024 May;56(3):382-391. doi: 10.1111/jnu.12959. Epub 2024 Jan 25. PMID 38273666